CLINICAL TRIAL: NCT05302037
Title: A Phase I Trial to Evaluate Allogeneic NKG2DL-targeting Chimeric Antigen Receptor-grafted γδ T Cells (CTM-N2D) in Subjects With Advanced Solid Tumours or Haematological Malignancies (the ANGELICA Trial)
Brief Title: Allogeneic NKG2DL-targeting CAR γδ T Cells (CTM-N2D) in Advanced Cancers (ANGELICA)
Acronym: ANGELICA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CytoMed Therapeutics Pte Ltd (Industry)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTM-N2D-102
Record Dates: First submitted 2022-03-20; First posted 2022-03-31 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Malignancy; Refractory Cancer; Relapsed Cancer
Keywords: cancer; malignancy; solid cancer; solid tumours; haematological cancer; haematological malignancy; refractory cancer; relapsed cancer; CAR-T; cell therapy; gamma delta
MeSH Terms: conditions — Neoplasms; Recurrence; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose-Escalation Arm (Experimental): Four infusions of CTM-N2D at escalating doses: 1x10^7, 1x10^8, 3x10^8 or 1x10^9 per infusion at an interval of one infusion every 7 days.
  Interventions: Biological: Allogeneic NKG2DL-targeting Chimeric Antigen Receptor-grafted γδ T Cells (CTM-N2D)
- Optimal Dose Arm (Experimental): Four infusions of CTM-N2D at the optimal dose (expected to be 1x10^9) at an interval of one infusion every 7 days.
  Interventions: Biological: Allogeneic NKG2DL-targeting Chimeric Antigen Receptor-grafted γδ T Cells (CTM-N2D)

INTERVENTIONS:
Biological: Allogeneic NKG2DL-targeting Chimeric Antigen Receptor-grafted γδ T Cells (CTM-N2D) — In the production of CTM-N2D, blood cells from healthy donors are used as starting materials. Through a proprietary expansion technology, γδ T cells of high-purity can be obtained. These γδ T cells are further grafted with NKG2DL-targeting CARs using mRNA electroporation to enhance its anticancer potency. The finished product (CTM-N2D) are then infused allogeneically into cancer patients.

SUMMARY:
CAR-T is a pioneering cancer treatment which has found success in some cancers. This treatment is made first by taking blood cells from the patient. Then in the lab, an artificial protein - a Chimeric Antigen Receptor (CAR), is grafted on the surface of immune cells. The modified cells, which are readministered to the patient, have enhanced abilities to target and destroy cancers than unmodified immune cells.

Currently approved CAR-T can only be used autologously. i.e. the patient will receive CAR-T treatment made from their own cells. This is because current CAR-T treatment uses αβ T cells - a type of immune cell which are largely non-transferable between individual human beings due to the high risk of Graft-versus-Host Disease. However, autologous CAR-T comes with many limitations. A lengthy, manufacturing process follows after the patient donates their own blood, accompanied by a high risk of manufacturing failure, which can be attributed to the cell quality from cancer patients undergoing stressful anti-cancer therapy.

CytoMed Therapeutics pioneers a new CAR-T treatment (CTM-N2D) which may confer some benefit over current CAR-T treatment. CTM-N2D uses a subtype of immune cell -- γδ T cell. Secondly, the CAR on CTM-N2D targets a surface antigen called NKG2DL which are commonly present in many cancer. These two features may confer a safer product profile, of better quality and may be efficacious in cancers where previous CAR-T treatments has not.

The phase I clinical trial of CTM-N2D will be conducted at the National University Hospital, Singapore. The objective of this clinical trial is to determine the optimal dose of CTM-N2D, and to investigate its safety and tolerability. The subjects of the clinical trial will also be investigated for their tumour response to CTM-N2D.

CTM-N2D has undergone preclinical studies. Relevant data from other clinical trials are also used to infer the expected outcome, and strategies of management of this clinical trial. The institution's ethical review board must give its approval before the study may begin. An independent Data Safety Monitoring Board monitors the safety aspect of this trial.

DETAILED DESCRIPTION:
Study Drug

The study treatment uses allogeneic NKG2DL-targeting CAR-grafted γδ T cells (also known as CTM-N2D). The treatment a) targets multiple stressed-induced cancer antigens (via the built-in receptors on γδ T cells, e.g., γδ TCR, NKG2D, DNAM-1); and (b) targets eight known NKG2DLs e.g., MICA/B, ULBP1-6 (via the grafted NKG2DL-targeting CAR). In humans, NKG2DLs are identified as MICA/B and ULBP1-6. Many tumour cell lines and primary tumours of various tissue-origins express NKG2DLs, providing attractive targets for CTM-N2D therapy

CTM-N2D refers to allogeneic γδ T cells that express CARs containing an extracellular domain of NKG2D as binding unit. CTM-N2D is manufactured from peripheral blood mononuclear cells (PBMCs) of allogeneic healthy donors through γδ T cell expansion and mRNA electroporation.

CTM-N2D will be packaged in an infusion bag to contain up to 1x10^9 cells in 100ml of infusible solution (saline with 5% human serum albumin) and delivered to the clinical site on the day of planned infusion. The transportation temperature will be maintained at 2 - 8°C.

Study Design

This is a two-cohort phase I study. In cohort 1 (interpatient dose-escalation cohort), the subjects will be given four infusions of CTM-N2D at escalating doses: 1x10^7, 1x10^8, 3x10^8 or 1x10^9 per infusion at an interval of one infusion every 7 days. This is to discern an optimal dose. In cohort 2 (optimal dose cohort), the subjects will be given four infusions of CTM-N2D at the optimal dose, which are given at an interval of one infusion every 7 days. This is to further confirm safety and tolerability.

If no DLT is detected in the first 3 patients in cohort 1, recruitment for cohort 2 will commence, with 6 patients to be treated with four doses of CTM-N2D at 1x10^9/infusion.

Patients in the interpatient dose-escalation cohort will be treated in sequence for the first four doses (i.e., only after all first four doses are administered for the first patient, will therapy for the second patient be allowed to commence). Such restriction is not extended to the maintenance doses. In the optimal dose cohort, 3 patients will be recruited, treated, and observed for DLT first, before another 3 patients are recruited. If 0/6 or 1/6 DLT is seen in the optimal dose cohort, the optimal dose will be established as RP2D.

If the patients do not demonstrate progressive disease after the first 4 doses of CTM-N2D and after the first imaging at 2 months from the start of study treatment (i.e., C1:1D1), maintenance doses of CTM-N2D will be manufactured and administered once every 2 months for a maximum of 5 doses. A computed tomography (CT) scan (or other forms of radiological assessment deemed appropriate by the investigator) will be performed every 2 months to evaluate stability (or response) of disease before manufacturing (a 20-day process) and administering each maintenance dose.

Treatment with CTM-N2D beyond 5 maintenance doses will be contingent to discussion with Sponsor and PI. Treatments with maintenance doses of CTM-N2D will not be considered in determining DLT.

Study Procedures and Assessments

Once informed consent is obtained and subject eligibility is confirmed, CytoMed will schedule and plan the manufacturing of CTM-N2D for the given subject.

The treatment regimen begins with lymphodepletion using Fludarabine and Cyclophosphamide to precondition the patient before the first treatment cycle with four weekly doses of CTM-N2D. Zoledronic acid will be given one day before each CTM-N2D infusion to maximize the potency of CTM-N2D.mTrial subjects will receive CTM-N2D by i.v infusion. To further enhance the survival of CTM-N2D, a dose of 1x10^6 IU/m2 IL-2 will be injected subcutaneously within 2 hours after each CTM-N2D infusion.

Clinical assessments will be performed at specified timepoints as written in the protocol. Any other relevant laboratory/imaging evaluations can be performed at any point in time, as deemed appropriate by the site investigator(s).

To assess patient well-being after CTM-N2D infusion as well as to monitor the pharmacokinetics and bioactivities of CTM-N2D, blood samples will be collected from trial subjects at various time points throughout the study period. Other blood investigations are to be performed at the clinical site as scheduled in the trial protocol and according to institutional guidelines. Additional laboratory investigations may be performed at the discretion of the investigator.

Assessments of tumour at specified timepoints, and are to be reported by a dedicated, independent radiologist, in accordance with RECIST criteria version 1.1. Other imaging modalities may be considered at the discretion of the investigator.

Off-study Follow-up and Assessments

In the event CTM-N2D therapy is discontinued due to PD or unacceptable AE, off-study follow-up and assessments will be performed up to 14 days from the date the subject is removed from the study.

If the trial subject is removed from the study due to unacceptable AE, the AE should be followed for at least 28 days from the last dose of study treatment until the AE is stabilized, or until the initiation of other anti-tumour therapy as off-study treatment, whichever comes first.

Post-study Follow-up and Procedures

Trial subjects will be followed for survival status, at the discretion of the investigator, from the end of the study until their death, or for a period of up to 48 months after the last patient was initiated for study treatment, whichever occurs first.

Discontinuation Visit and Procedures

Upon voluntary withdrawal from the study, trial subject will still be given the option to continue scheduled evaluations, as well as, to complete an end of study evaluation. Appropriate medical care will continue to be meted out by the clinicians at the study site.

Safety, Adverse Events and Toxicity Management

Safety of the study treatment regimen will be assessed by monitoring and recording any toxicities or Aes appeared in trial subjects during the study period. The descriptions of Aes and their grading scales found in the NCI CTCAE v5.0 will be utilized for AE reporting.

Reporting of Events

The investigator is expected to collect, record, and report the "Unanticipated Problems Involving Risk to Subjects or Others" ("UPIRTSO") events in the study to the NHG Domain Specific Review Boards (DSRB). The criteria for UPIRTSO events and their timeline for reporting to NHG DSRB are defined in the protocol.

Reporting of SAEs to HSA

The investigator is expected to collect, record and report SAEs to the Health Science Authority (HSA) through CytoMed Therapeutics Pte Ltd. All SAEs that are unexpected and related to the study drug will be reported to HSA.

All SAEs that are unexpected and related to the study drug will be reported. The investigator is responsible for informing CytoMed Therapeutics Pte Ltd within 24 hours after first knowledge that the case qualifies for expedited reporting. CytoMed Therapeutics Pte Ltd will report the SAEs to HSA no later than 15 calendar days upon receiving SAE reports from the investigator. Follow-information will be actively sought and submitted as it becomes available. For fatal or life-threatening cases, HSA will be notified as soon as possible but no later than 7 calendar days after first knowledge that a case qualifies, followed by a complete report within 8 additional calendar days.

Safety Monitoring Plan

The investigator is responsible for appropriate medical care of subjects during the study. The investigator will review all patients to monitor toxicity before each treatment cycle. If a subject reports an AE, appropriate care and follow-up evaluation should be implemented by the investigator until the event is either resolved or stable.

An independent Data Safety Monitoring Board (iDSMB) formed by experts with relevant knowledge of the study will monitor the safety aspect of this trial. The board will review the safety data after completion of each cohort and/or if a DLT occurs.

Dose-limiting Toxicities (DLTs)

DLT is defined as an unexpected grade 3 or 4 non-hematologic toxicity that is probably related to CTM-N2D infusion and experienced within 8 weeks immediately after the start of study treatment (i.e., C1:1D1). Treatments with maintenance doses of CTM-N2D will not be considered in determining DLT. The criteria for DLT is defined in the protocol.

Whenever a patient experiences toxicity that fulfil the criteria for a DLT, the study treatment will be interrupted. The investigator is responsible for reporting DLT observed by the investigator to the sponsor within 24 hours of learning of its occurrence.

Toxicity Management

Current CAR-T cell therapy has been used to treat B-cell malignancies and multiple myeloma. The clinical experiences from these trials show that potential severe toxicities are not uncommon. Such potential severe toxicities in CAR-T therapy include cytokine release syndrome (CRS), immune effector cell-associated neurotoxicity syndrome (ICANS), on-target off-tumour toxicity, tumour lysis syndrome (TLS) and immunogenicity.

The grading and management of potential CAR-T toxicities follow a grading system proposed by the American Society for Transplantation and Cellular Therapy (ASTCT; formerly American Society for Blood and Marrow Transplantation, ASBMT). However, institution practices and sub-specialty input will prevail and supersede this protocol if necessary.

A specific concern for CTM-N2D treatment is the potential "on-target off-cancer" toxicity. CTM-N2D targets NKG2D ligands, which may be upregulated in non-cancer cells upon infection, inflammation, or stress. The recognition of the non-cancer cells by CTM-N2D may cause CRS and autoimmune toxicity. Subjects will also monitored for Tumour lysis syndrome (TLS).

Subject Withdrawal

Subjects have the right to withdraw from the study at any time and for any reason, without prejudice to their future medical care by the investigator or at the institution. Subjects who do not complete the study protocol will be considered to have prematurely discontinued study. The reasons for premature discontinuation (for example, voluntary withdrawal, toxicity, death) must be recorded on the case report form. Final study evaluations will be completed at the time of discontinuation.

The investigator and/or sponsor can also decide to withdraw a subject from the investigational product and/or other protocol-required therapies, protocol procedures, or the study as a whole or at any time prior to study completion.

Study Monitoring

The principal investigator is responsible for familiarising the investigator(s) and the entire study team involved in the study with all study procedures, including the administration of the study drug. The investigators are responsible for monitoring the safety of subjects who have enrolled for this study and for alerting the principal investigator to any event that seems unusual, even if this event may be considered an unanticipated benefit to the subject. The investigators are responsible for appropriate medical care of subjects throughout the study period.

In the event of SAEs, or Aes that result in any subject(s) withdrawing from the study, the investigators remain responsible for the care and followup of the subject(s), until the AE resolves, stabilizes or is explained.

Data collection and analysis

Data are recorded and stored on an electronic data capturing system called Redcap. CRFs will be translated to SPSS and Excel spreadsheets for further analysis. ANOVA multivariate analysis will be used to determine statistical significance of continuous variables. Chi-square and Fisher's exact test will be used to assess associations between categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age
* Provision of signed and dated, written informed consent prior to any study specific procedures, sampling, and analyses (if applicable, the written informed consent may include access to all archival tumour tissue, e.g., diagnostic and/or most recent samples for correlative study)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 and an estimated life expectancy of greater than 12 weeks
* Females of reproductive age group must be on effective contraception (if sexually active), must not be breast feeding and must have a negative pregnancy test prior to the start of lymphodepletion.
* For the duration of the study and for 1 week after the last study drug administration, sexually active male patients must be willing to use barrier contraception (i.e., condoms) with all sexual partners. Where the sexual partner is a 'woman of child-bearing potential' who is not using effective contraception, the male patients must use a condom (with spermicide) during the study and for 6 months after the last dose of a study drug.
* Adequate hepatic, renal and lung function as demonstrated by any of the following laboratory values:

  * AST or ALT ≤ 3 x ULN
  * Total bilirubin ≤ 1.5 x ULN
  * Glomerular filtration rate (GFR) > 50 mL/min, as assessed using the Cockroft-Gault formula or 24 h urine creatinine collection
  * SpO2 on room air > 94%
* Adequate bone marrow reserve as demonstrated by any of the following laboratory values:

  * Absolute neutrophil count (ANC) ≥ 1.0x10^9/L
  * Platelet count ≥ 75 x 10^9/L
  * Haemoglobin ≥ 9.0 g/dL
* Patients must have a metastatic cancer resistant to or deemed unsuitable for at least two standard lines of cancer therapy regimens, as part of their management of recurrent/persistent disease.
* Presence of measurable tumour by RECIST 1.1 criteria
* Serum 25 Hydroxyvitamin D total ≥ 20ng/ml
* Have a diagnosis of cancer that is known to express NKG2D ligands

Exclusion Criteria:

* With the exception of alopecia, any unresolved toxicities from prior therapy ≥ the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grade 2
* Spinal cord compression or brain metastases unless asymptomatic, stable and not requiring steroids for at least 4 weeks prior to the start of lymphodepletion
* As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, active bleeding diatheses, renal transplant, or active infection including any patient known to have human immunodeficiency virus (HIV) or hepatitis virus. Screening for chronic conditions is not required.
* All HBsAg-positive patients (For HBsAg-negative, but anti-HBc total-positive patients, HBV viral load will be further tested. If HBV viral load is negative, patients may be included.)
* Active or prior documented autoimmune or inflammatory disorders including inflammatory bowel disease (e.g., colitis or Crohn's disease), diverticulitis (with the exception of diverticulosis), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc). The following are exceptions to this criterion:

  * Subjects with vitiligo or alopecia
  * Subjects with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Subjects without active disease in the last 5 years may be included but only after consultation with the medical monitor
  * Subjects with celiac disease controlled by diet alone
  * For other autoimmune or inflammatory conditions not specifically mentioned, discuss on case-by-case basis with investigator and medical monitor
* Concurrent severe and/or uncontrolled medical condition (e.g., severe COPD, severe Parkinson's disease, active inflammatory bowel disease) or psychiatric condition (screening for chronic disease is not required)
* Female patients who are breast-feeding or patients of reproductive potential who are not employing an effective method of contraception
* Receiving, or having received during the four weeks prior the start of lymphodepletion, any investigational product
* Treatment with any investigational biological product (e.g., immune check point blockers, antibodies, nanoparticles, experimental) during the four weeks prior the start of lymphodepletion
* Patients who underwent major surgery during the four weeks prior to the start of lymphodepletion
* Radiation (except planned or ongoing palliative radiation to bone outside of the region of measurable disease) during the three weeks prior to the start of Lymphodepletion
* Active infection requiring systemic long-term (> 2 weeks) treatment with antibiotics, antifungal or antiviral drugs
* Cardiac dysfunction as defined as: Myocardial infarction within six months of study entry, NYHA Class II/III/IV heart failure, unstable angina, unstable cardiac arrhythmias or reduced LVEF < 50%.
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTc) > 470 msec
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block)
  * Uncontrolled hypertension requiring clinical intervention
* Failed dental clearance (for zoledronic acid administration)
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements

Subject Withdrawal Criteria

Treatment may continue until one of the following criteria applies:

* Disease progression
* Intercurrent illness that prevents further administration of treatment
* Unacceptable adverse event(s)
* Intolerable non-hematologic toxicities ≥ NCI CTCAE v5.0 Grade 2
* Unmanageable hematologic or non-hematologic toxicities ≥ NCI CTCAE v5.0 Grade 3
* General or specific changes in the patient's condition that renders the patient unsuitable for further treatment at the discretion of the investigator
* Patient who cannot recover from adverse event(s) and lead to treatment delay for > 4 weeks
* Patient who decides to withdraw from the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To determine a dose regimen and schedule of CTM-N2D at which no more than one patient out of up to six patients at the same dose level experience a CTM-N2D-related DLT | Within 8 weeks immediately after the start of study treatment
  Cohort 1: Three patients will be treated with four escalating doses of CTM-N2D to determine an optimal dose based on the incidence of DLT. DLT is defined as an unexpected grade 3 or 4 non-hematologic toxicity that is probably related to CTMN2D infusion and experienced within 8 weeks immediately after the start of study treatment. Treatments with maintenance doses of CTM-N2D will not be considered in determining DLT.
Number of Participants With Treatment-Related Adverse Events as assessed by NCI CTCAE v5.0 | 24 months after the start of study treatment
  Cohort 2: Six patients will be treated with four infusions of CTM-N2D at the optimal dose determined in Cohort 1.

SECONDARY OUTCOMES:
Maximum objective response rate according to RECIST v1.1 | 24 months after the start of study treatment
  Tumour Asessments
Progression-free survival (PFS) | Up to 48 months after the last patient was initiated for study treatment
  Trial subjects will be followed for survival status, at the discretion of the investigator, from the end of the study until their death, or for a period of up to 48 months after the last patient was initiated for study treatment, whichever occurs first.
Overall survival (OS) | Up to 48 months after the last patient was initiated for study treatment
  Trial subjects will be followed for survival status, at the discretion of the investigator, from the end of the study until their death, or for a period of up to 48 months after the last patient was initiated for study treatment, whichever occurs first.
Duration of response in patients with objective response up to M24 after the start of study treatment (i.e., C1:1D1) | Up to 48 months after the last patient was initiated for study treatment
  Trial subjects will be followed for survival status, at the discretion of the investigator, from the end of the study until their death, or for a period of up to 48 months after the last patient was initiated for study treatment, whichever occurs first.

OTHER OUTCOMES:
Detection and quantification of lymphocyte subsets including γδ T cell subset in blood | 24 months after the start of study treatment
  CTM-N2D related blood test
Detection and quantification of serum cytokines | 24 months after the start of study treatment
  CTM-N2D related blood test

CONTACTS AND LOCATIONS:
Overall Officials: Anand D Jeyasekharan, Dr, Principal Investigator — National University Health System (NUHS); Jieming Zeng, Dr, Study Director — CytoMed Therapeutics Pte Ltd
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demoulin B, Cook WJ, Murad J, Graber DJ, Sentman ML, Lonez C, Gilham DE, Sentman CL, Agaugue S. Exploiting natural killer group 2D receptors for CAR T-cell therapy. Future Oncol. 2017 Aug;13(18):1593-1605. doi: 10.2217/fon-2017-0102. Epub 2017 Jun 14. PMID 28613086
- [Background] Nakajima J, Murakawa T, Fukami T, Goto S, Kaneko T, Yoshida Y, Takamoto S, Kakimi K. A phase I study of adoptive immunotherapy for recurrent non-small-cell lung cancer patients with autologous gammadelta T cells. Eur J Cardiothorac Surg. 2010 May;37(5):1191-7. doi: 10.1016/j.ejcts.2009.11.051. PMID 20137969
- [Background] Wada I, Matsushita H, Noji S, Mori K, Yamashita H, Nomura S, Shimizu N, Seto Y, Kakimi K. Intraperitoneal injection of in vitro expanded Vgamma9Vdelta2 T cells together with zoledronate for the treatment of malignant ascites due to gastric cancer. Cancer Med. 2014 Apr;3(2):362-75. doi: 10.1002/cam4.196. Epub 2014 Feb 7. PMID 24515916
- [Background] Wilhelm M, Smetak M, Schaefer-Eckart K, Kimmel B, Birkmann J, Einsele H, Kunzmann V. Successful adoptive transfer and in vivo expansion of haploidentical gammadelta T cells. J Transl Med. 2014 Feb 15;12:45. doi: 10.1186/1479-5876-12-45. PMID 24528541
- [Background] Neelapu SS. Managing the toxicities of CAR T-cell therapy. Hematol Oncol. 2019 Jun;37 Suppl 1:48-52. doi: 10.1002/hon.2595. PMID 31187535
- [Background] Neelapu SS, Tummala S, Kebriaei P, Wierda W, Gutierrez C, Locke FL, Komanduri KV, Lin Y, Jain N, Daver N, Westin J, Gulbis AM, Loghin ME, de Groot JF, Adkins S, Davis SE, Rezvani K, Hwu P, Shpall EJ. Chimeric antigen receptor T-cell therapy - assessment and management of toxicities. Nat Rev Clin Oncol. 2018 Jan;15(1):47-62. doi: 10.1038/nrclinonc.2017.148. Epub 2017 Sep 19. PMID 28925994